CLINICAL TRIAL: NCT01171612
Title: Evaluation and Monitoring of Perioperative Management of Patients With Coronary Stents Undergoing Noncardiac Surgery
Brief Title: Perioperative Management of Patients With Coronary Stents Undergoing Noncardiac Surgery
Acronym: RegistStents
Status: Completed | Type: Observational
Sponsor: Corporacion Parc Tauli (Other)
Responsible Party: Principal Investigator, Anna Rodriguez Pont, MD, Corporacion Parc Tauli
Other Study IDs: CIR2009017
Record Dates: First submitted 2010-07-23; First posted 2010-07-28 (Estimated); Results first posted 2013-11-25 (Estimated); Last update posted 2016-04-07 (Estimated); Status verified 2016-03

CONDITIONS: Acute Coronary Syndrome; Coronary Stent Occlusion; Surgery
Keywords: Coronary Stent; BMS stent; DES stent; Date of stent implantation; cardiac event; neurovascular event; Bleeding; transfusion
MeSH Terms: conditions — Acute Coronary Syndrome; Cardiovascular Diseases; Hemorrhage

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Coronary Stent: Patients with coronary Bare Metal Stent (BMS) or Drug Eluting Stent (DES) undergoing noncardiac surgery

SUMMARY:
The purpose of this study is to evaluate and monitor perioperative management of patients with coronary stents undergoing noncardiac surgery.

Objectives:

* To describe the incidence and severity of adverse cardiovascular events in patients with coronary stents undergoing noncardiac surgery with admission.
* To assess the following-up of the guidelines about the perioperative management of antiplatelet therapy in these patients.
* To assess the relationship between the incidence of cardiac or neurovascular events, as well as bleeding complications with the perioperative management of antiplatelet therapy.
* Number of Participants with Adverse Events as a Measure of Safety

DETAILED DESCRIPTION:
(Not desired)

ELIGIBILITY:
Inclusion Criteria:

* > 18 years old, with coronary stents
* American Society of Anaesthesia physical status II-V
* noncardiac surgery wiht admission
* informed consent

Exclusion Criteria:

* < 18 years old
* American Society of Anaesthesia physical status I
* ambulatory surgery
* pregnancy
* obstetric anaesthesia
* endoscopic procedures
* cardiac surgery
* not informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with coronary stents undergoing noncardiac surgery with admission between May 2010 and April 2012
Sampling Method: Non-Probability Sample
Enrollment: 483 (Actual)
Dates: Start 2009-06; Primary Completion 2010-02 (Actual); Study Completion 2012-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Anna Rodriguez-Pont, MD, Principal Investigator — Corporacio Sanitaria Parc Tauli
Locations (13):
- Spain (13):
  - Hospital Germans Trias i Pujol, Badalona, Barcelona
  - Hospital Municipal de Badalona, Badalona, Barcelona
  - Fundació Puigvert - IUNA, Barcelona, Barcelona
  - Hospital Clínic, Barcelona, Barcelona
  - Parc de Salut Mar-Esperança, Barcelona, Barcelona
  - Parc de Salut Mar, Barcelona, Barcelona
  - Hospital Igualada, Igualada, Barcelona
  - Hospital de Mataró, Mataró, Barcelona
  - Hospital de Sabadell. Corporació Sanitària Parc Taulí, Sabadell, Barcelona
  - Hospital de Sant Celoni, Sant Celoni, Barcelona
  - Clínica ASEPEYO, Sant Cugat del Vallès, Barcelona
  - Hospital Sant Joan Despi Moisès Broggi, Sant Joan Despí, Barcelona
  - Hospital Mútua de Terrassa, Terrassa, Barcelona

REFERENCES:
- [Derived] Rodriguez A, Guilera N, Mases A, Sierra P, Oliva JC, Colilles C; REGISTRESTENTS group. Management of antiplatelet therapy in patients with coronary stents undergoing noncardiac surgery: association with adverse events. Br J Anaesth. 2018 Jan;120(1):67-76. doi: 10.1016/j.bja.2017.11.012. Epub 2017 Nov 21. PMID 29397139

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Observational, multicenter and prospective study, approved by the Ethics Committee. All patients with coronary stents undergoing noncardiac surgery with admission from February 2010 to April 2012 were the basis of the study.
Pre-assignment Details: Patients scheduled for noncardiac surgery with admission
Period: Overall Study
Arm/Group | Coronary Stent
Started | 483
Completed | 432
Not Completed | 51
Not completed — Lost to Follow-up | 51

BASELINE CHARACTERISTICS:
Population: 20 patienet were not taking previous antiplatelet agents
Arm/Group | Coronary Stent
Number analyzed (Participants) | 432
Age, Customized [Number; unit: participants] — age < or = 70 years old age > 70 years old
  participants
    Between 18 and 70 years | 219
    >70 years | 213
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 72
  Male | 360
Region of Enrollment [Number; unit: participants]
  Spain | 432
Body Mass Index [Median (Full Range); unit: Kgm^2] | 27.9 [18.0 to 50.0]
Antiplatelet Therapy [Number; unit: participants] — patients taking previous aspirin, clopidogrel or both
  participants
    Antiplatelet therapy | 412
    Not antiplatelet therapy | 20

OUTCOME MEASURES:

1. Primary Outcome: Major Adverse Cardiac and Cerebrovascular Events (MACCEs)
Description: Cardiac Mortality, Myocardial Infarction, Angina Pectoris, new arrythmia, Congestive Heart Failure, Stroke, Cardiac Arrest
Time Frame: up to 90 days after surgery
Measure: Number; unit: participants
Arm/Group | Coronary Stent
Number analyzed (Participants) | 432
participants | 63

2. Secondary Outcome: Major Haemorrhagic Events
Description: Transfusion > = 2 red blood cells Units, haemoglobin descent >= 20 gr/dL, intracerebral haemorrhage
Time Frame: up to 90 days after surgery
Measure: Number; unit: participants
Arm/Group | Coronary Stent
Number analyzed (Participants) | 432
participants | 161

3. Secondary Outcome: Number of Patients With Adverse Events Related With Antiplatelet Therapy Management
Description: Perioperative withdrawal antiplatelet therapy is defined with > or = 5 days without therapy
  We create 3 categories:
  1. Not withdrawal
  2. Complete withdrawal (5 or > days without antiplatelet drugs , mono or dual therapy)
  3. Incomplete withdrawal: patients under dual antiplatelet therapy, who maintain aspirin and stopped clopidogrel =/ > 5 days
Time Frame: 90 days after surgery
Population: MACCEs
Measure: Number; unit: participants
Groups:
- Not Withdrawal Antiplatelet Therapy: Patients wiht aspirin and/or clopidogrel withdrawal for 5 or more days
- Incomplete Withdrawal (Mantaining ASA, Clopidogrel Withdrawn): Patients under dual antiplatelet therapy, wich maintain aspirin, and withdrawn clopidogrel 5 or more days
- Complete Withdrawal: patients with aspirin oand/or clopidogrel, which stopped therapy > 5 days
Arm/Group | Not Withdrawal Antiplatelet Therapy | Incomplete Withdrawal (Mantaining ASA, Clopidogrel Withdrawn) | Complete Withdrawal
Number analyzed (Participants) | 294 | 72 | 46
participants | 38 [0.733 to 3.662] | 10 [0.513 to 2.299] | 9
Statistical Analysis 1: Comparison: Not Withdrawal Antiplatelet Therapy vs Incomplete Withdrawal (Mantaining ASA, Clopidogrel Withdrawn); Reference group were patients who maintained antiplatelet drugs (aspirin and/or clopidogrel) during the 4 days before surgery; Test type: Superiority or Other; p = 0.479, Chi-squared; Odds Ratio (OR) = 1.086, 95% CI 2-sided [0.513 to 2.299]
Statistical Analysis 2: Comparison: Not Withdrawal Antiplatelet Therapy vs Complete Withdrawal; Test type: Superiority or Other; p = 0.479, Chi-squared; Odds Ratio (OR) = 1.638, 95% CI 2-sided [0.733 to 3.662]

ADVERSE EVENTS:
Time Frame: Perioperative events from surgery to 90 days after
Description: We registered the adverse events from surgery to 90 days after All the events were included in our outcomes definitions
Groups:
- Cardiac and Cerebrovascular Events: Adverse events registered independently related with antiplatelet therapy management
Arm/Group | Cardiac and Cerebrovascular Events
Serious Adverse Events (participants affected / at risk) | 61/432
Other Adverse Events (participants affected / at risk) | 6/432
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cardiac and Cerebrovascular Events (N=432)
Cardiac Arrest (Cardiac disorders) | 1 (1) — In hospital Cardiac arrest
Cardiac Death (Cardiac disorders) | 1 (1) — Death with cardiac origin
Acute Myocardial Infarction (Cardiac disorders) | 12 (13)
Unstable Angina (Cardiac disorders) | 39 (39)
Significant Arrythmia (Cardiac disorders) | 13 (15)
Cardiac Failure (Cardiac disorders) | 8 (8)
OTHER ADVERSE EVENTS (reported when occurring in more than 0.2% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cardiac and Cerebrovascular Events (N=432)
Stroke, Transient Ischaemic Attack (Nervous system disorders) | 4 (4)
Deep Venous Thrombosis (Vascular disorders) | 1 (1)
Arterial ischaemia (Vascular disorders) | 1 (1)

LIMITATIONS AND CAVEATS:
This is a prospective and observational study

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes